CLINICAL TRIAL: NCT03519477
Title: A Pilot Prospective, Randomized Controlled Trial Assessing the Impact of Clinical Decision Support Using Comprehensive Medication Monitoring on Heart Failure Patient Outcomes
Brief Title: Comprehensive Medication Monitoring on Heart Failure Patient Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated by sponsor for commercial reasons
Sponsor: Precera Bioscience, Inc. (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SAN_UPMC_CV_001
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure，Congestive
Keywords: clinical decision support; drug levels in blood; therapeutic drug monitoring; medication adherence; medication therapy management
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart failure care with Sano test (Experimental): Scheduled outpatient care for patients at high risk of admission for heart failure, supplemented with the Sano Patient Medication Profile
  Interventions: Diagnostic Test: Sano Patient Medication Profile
- Heart failure care as-usual (No Intervention): Scheduled outpatient care for patients at high risk of admission for heart failure, care as-usual (i.e. without the Sano Patient Medication Profile).

INTERVENTIONS:
Diagnostic Test: Sano Patient Medication Profile — The Sano Patient Medication Profile (PMP) is a graphical report comparing prescribed medications to liquid (chromatography/tandem mass-spectrometry) LC/MS/MS-detected drugs from patient blood samples
  Arms: Heart failure care with Sano test

SUMMARY:
The purpose of this study is to evaluate the clinical utility of comprehensive medication monitoring using the Patient Medication Profile to improve heart failure patient medication therapy and associated outcomes relative to usual care in a hospital setting.

DETAILED DESCRIPTION:
Congestive heart failure has an exceptionally high rate of hospital admission and is responsible for more re-admissions (23.5% at 30 days) in the United States than the 2nd and 3rd leading causes combined. Inadequate medication reconciliation both on admission and discharge from the hospital is a significant cause of medical error. In one study of cardiovascular patients, 44% believed they were taking a medication they were not, and 96% were unable to recall at least one medication they were taking. In the same study patients omitted on average 6.8 medications from their medication list. Medication optimization through improved adherence and reconciled medical records has been postulated to significantly improve admission and 30-day hospital readmission rates.

Sano has developed a blood-based comprehensive medication monitoring tool that identifies and quantitates 235 prescription drugs and drug metabolites. It does not detect illicit drugs. This tool, which produces an output report designated the 'Patient Medication Profile', is designed to be used with clinical decision support to improve medication adherence, reduce medication errors, and optimize medication therapy. For heart failure patients, the investigators hypothesize that deploying the Patient Medication Profile with clinical decision support at key points of treatment intervention will A) improve medication adherence, B) identify and reconcile significant discrepancies in the medication list, C) result in reduced hospital admissions, and D) result in better overall patient outcomes. These outcome expectations are relative to usual care for heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a regularly scheduled visit to a University of Pittsburgh Medical Center (UPMC) cardiology clinic in Oakland
* Patients must have Heart Failure with Reduced Ejection Fraction (≤40%)
* Patients have admitted to UPMC hospital facility between one and five times in past 12 months
* Patients must be able to provide informed consent for present study
* Patient age > 18 years

Exclusion Criteria:

* Enrolled in Hospice
* Patient on home inotrope (Dobutamine or milrinone)
* World Health Organization (WHO) Group 1 or Group 5 pulmonary hypertension
* Patient with current ventricular assist device (VAD)
* Not able to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Change in adherence to prescribed cardiology medications | 30 days
  For each patient, the proportion of prescribed medications that are detected using the baseline and final PMP will be calculated; change in adherence will be defined as proportion using final PMP, minus proportion using baseline PMP. Compare adherence difference in intervention vs. control groups.

SECONDARY OUTCOMES:
Number of hospital admissions per patient within 90 days of enrollment in intervention vs. control group | 90 days
Baseline adherence to prescribed cardiology medications as a predictor of hospital admission for heart failure within 90 days | 90 days
  Baseline adherence to prescribed cardiology medications as a predictor of hospital admission for heart failure within 90 days. This endpoint will use baseline adherence and the Patient Medication Profile will not have been discussed with the care team in the intervention group, therefore both intervention and control groups will be pooled
Drug Related Problem identification and resolution | 30 days
  Documented drug related problems identified by medication reconciliation will be compared between the intervention and control groups. The number of changes in medications to resolve drug related problems, such as medication additions, terminations, dosage or frequency changes will be compared between the intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Heart and Vascular Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cumbler E, Wald H, Kutner J. Lack of patient knowledge regarding hospital medications. J Hosp Med. 2010 Feb;5(2):83-6. doi: 10.1002/jhm.566. PMID 20013875
- [Background] Gupta P, Patel P, Strauch B, Lai FY, Akbarov A, Maresova V, White CMJ, Petrak O, Gulsin GS, Patel V, Rosa J, Cole R, Zelinka T, Holaj R, Kinnell A, Smith PR, Thompson JR, Squire I, Widimsky J Jr, Samani NJ, Williams B, Tomaszewski M. Risk Factors for Nonadherence to Antihypertensive Treatment. Hypertension. 2017 Jun;69(6):1113-1120. doi: 10.1161/HYPERTENSIONAHA.116.08729. Epub 2017 May 1. PMID 28461599